CLINICAL TRIAL: NCT05786716
Title: DETERMINE (Determining Extended Therapeutic Indications for Existing Drugs in Rare Molecularly Defined Indications Using a National Evaluation Platform Trial): An Umbrella-Basket Platform Trial to Evaluate the Efficacy of Targeted Therapies in Rare Adult, Paediatric and Teenage/Young Adult (TYA) Cancers With Actionable Genomic Alterations, Including Common Cancers With Rare Actionable Alterations. Treatment Arm 04: Trastuzumab in Combination With Pertuzumab in Adult, Paediatric and Teenage/Young Adult Patients With Cancers With HER2 Amplification or Activating Mutations.
Brief Title: DETERMINE Trial Treatment Arm 04: Trastuzumab in Combination With Pertuzumab in Adult, Paediatric and Teenage/Young Adult Patients With Cancers With HER2 Amplification or Activating Mutations
Acronym: DETERMINE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: University of Manchester (Other); University of Birmingham (Other); Royal Marsden NHS Foundation Trust (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/21/004 - Treatment Arm 4; IRAS ID: 1004057 (Other: IRAS)
Record Dates: First submitted 2023-02-22; First posted 2023-03-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Haematological Malignancy; Colorectal Neoplasms; Urinary Bladder Neoplasm; Gallbladder Neoplasms; Salivary Gland Neoplasm; Lung Neoplasm; Pancreatic Neoplasm; Ovarian Neoplasms; Prostatic Neoplasm; Skin Neoplasm; Solid Tumour
Keywords: Adult; Antibodies, monoclonal; Cancer; Child; Molecular Targeted Therapy; Mutation; Paediatric; Pertuzumab; Precision Medicine; Rare; Receptor, ErbB-2; Targeted; Trastuzumab; Tumour-agnostic; Young adult
MeSH Terms: conditions — Hematologic Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms; Gallbladder Neoplasms; Salivary Gland Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Skin Neoplasms; Neoplasms | interventions — Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm 04: trastuzumab in combination with pertuzumab (Experimental): This trastuzumab and pertuzumab treatment arm is for adult, paediatric and TYA patients with cancers with HER2 amplification or activating mutations.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Trastuzumab — An initial loading dose of 8 mg/kg body weight, followed thereafter by a maintenance dose of 6 mg/kg body weight administered intravenously every 21 days. Patients may continue until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Herceptin
Drug: Pertuzumab — An initial loading dose of 640 mg, followed thereafter by a maintenance dose of 420 mg administered intravenously every 21 days. Paediatric patients will receive an initial loading dose of 14 mg/kg (maximum 840 mg), followed thereafter by a maintenance dose of 7 mg/kg (maximum 420 mg) administered intravenously every 21 days. Patients may continue until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Perjeta

SUMMARY:
This clinical trial is looking at a combination of drugs called trastuzumab and pertuzumab. This combination of drugs is approved together as standard of care treatment for adult patients with breast cancer (often with other anti-cancer drugs). This means it has gone through clinical trials and been approved by the Medicines and Healthcare products Regulatory Agency (MHRA) in the UK.

Trastuzumab and pertuzumab work in patients with these types of cancers which have a molecular alteration called HER2 amplification or HER2 activating mutation.

Investigators now wish to find out if it will be useful in treating patients with other cancer types which are also HER2 amplified or HER2 mutated. If the results are positive, the study team will work with the NHS and the Cancer Drugs Fund to see if these drugs can be routinely accessed for patients in the future.

This trial is part of a trial programme called DETERMINE. The programme will also look at other anti-cancer drugs in the same way, through matching the drug to rare cancer types or ones with specific mutations.

DETAILED DESCRIPTION:
DETERMINE Treatment Arm 04: Trastuzumab in combination with pertuzumab in Adult, Paediatric and TYA patients with rare* cancers with HER2 amplification or activating mutations and in common cancers where HER2 amplification or activating mutations are considered to be infrequent.

*Rare is defined generally as incidence less than 6 cases in 100,000 patients (includes paediatric and teenagers/young adult cancers) or common cancers with rare alterations.

This treatment arm has a target sample size of 30 evaluable patients. Sub-cohorts may be defined and further expanded to a target of 30 evaluable patients each.

The ultimate aim is to translate positive clinical findings to the NHS (Cancer Drugs Fund) to provide new treatment options for rare adult, paediatric and TYA cancers.

OUTLINE:

Pre-screening: The Molecular Tumour Board (MTB) makes a treatment recommendation for the patient based on molecularly-defined cohorts.

Screening: Consenting patients undergo biopsy and collection of blood samples for research purposes.

Treatment: Patients will receive trastuzumab and pertuzumab until disease progression without clinical benefit, unacceptable adverse events (AEs) or withdrawal of consent. Patients will also undergo collection of blood samples at various intervals while receiving treatment and at End of Treatment (EoT).

After completion of study treatment, patients are followed up every 3 months for 2 years.

THE DETERMINE TRIAL MASTER (SCREENING) PROTOCOL:

Please see DETERMINE Trial Master (Screening) Protocol record (NCT05722886) for information on the DETERMINE Trial Master Protocol and applicable documents.

ELIGIBILITY:
THE PATIENT MUST FULFIL THE ELIGIBILITY CRITERIA WITHIN THE DETERMINE MASTER PROTOCOL (NCT05722886) AND WITHIN THE TREATMENT ARM 04 (TRASTUZUMAB AND PERTUZUMAB) OUTLINED BELOW*

*When trastuzumab- and pertuzumab-specific inclusion/exclusion criteria or precautions below differ from those specified in the Master Protocol, the trastuzumab- and pertuzumab-specific criteria will take precedence.

Inclusion Criteria:

A. Confirmed diagnosis of a malignancy harbouring HER2 amplification, or an appropriate activating mutation as defined by the MTB, using an analytically validated next-generation sequencing method.

• A HER2 amplification copy number between 5-9 will require an MTB discussion. A HER2 amplification copy number ≥10 will be fast-tracked for an MTB recommendation, unless there are any patient-specific individualities (such as multiple gene amplifications) that require MTB discussion.

B. Age 12 years or above.

C. Women of childbearing potential are eligible provided that they meet the following criteria:

Have a negative serum or urine pregnancy test before enrolment and;

Agree to use one form of effective birth control method such as:

I. combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal):

II. progestogen-only hormonal contraception associated with or without inhibition of ovulation (oral, injectable or implantable)

III. intrauterine device (IUD)

IV. intrauterine hormone-releasing system (IUS)

V. bilateral tubal occlusion

VI. vasectomised partner

VII. sexual abstinence

VIII. male or female condom with or without spermicide

IX. cap, diaphragm or sponge with spermicide

Effective from the first administration of trastuzumab or pertuzumab (whichever is first), throughout the trial and for seven months after the last administration of trastuzumab or pertuzumab (whichever is later).

D. Male patients with partners who are women of childbearing potential are eligible provided that they agree to the following, from the first administration of trastuzumab or pertuzumab (whichever is first), throughout the trial and for seven months after the last administration of trastuzumab or pertuzumab (whichever is later):

* Agree to take measures not to father children by using a barrier method of contraception (condom plus spermicide) or to sexual abstinence.
* Non-vasectomised male patients with partners who are women of childbearing potential must also be willing to ensure that their partner uses an effective method of contraception as in C, above.
* Male patients with pregnant or lactating partners must be advised to use barrier method contraception (e.g. condom) to prevent drug exposure of the foetus or neonate.

All male patients must refrain from donating sperm for the same period.

E. Patients must be able and willing to undergo a fresh tissue biopsy at baseline and blood samples for translational research. Note that for patients with haematological malignancies or neuroblastomas, blood, bone marrow aspiration and/or trephine or lymph node biopsy samples may be taken.

F. ADULT PATIENTS (≥18 years): Adequate organ function as per haematological and biochemical indices within the ranges defined in the protocol. These measurements should be performed to confirm the patient's eligibility.

G. PAEDIATRIC PATIENTS (<18 years): Adequate organ function as per haematological and biochemical indices within the ranges defined in the protocol. These measurements should be performed to confirm the patient's eligibility.

Exclusion Criteria:

A. Diagnosis of HER2-positive early or metastatic breast cancer.

B. Female patients who are pregnant, breastfeeding or planning to become pregnant during the trial or within seven months following their last dose of trastuzumab or pertuzumab (whichever is later).

C. Severe dyspnoea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy.

D. Known hypersensitivity to trastuzumab or pertuzumab, murine proteins, or to any of the excipients.

E. Patients who were administered a live, attenuated vaccine within 28 days prior to enrolment, or anticipation of need for such a vaccine during trastuzumab and pertuzumab treatment or within six months after the final dose of trastuzumab and pertuzumab.

F. Patients with clinically significant pre-existing cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias (within three months), NYHA class III or IV congestive heart failure.

Left Ventricular Ejection Fraction <55%.

Patients with a cerebrovascular event (including stroke or transient ischaemic attack [TIA]) or cardiovascular event (including acute myocardial infarction [MI]) within three months before the first dose of trastuzumab and pertuzumab.

• Patients with primary CNS tumours may be considered unless intra-tumoural bleeding has occurred within 2 weeks of the first dose of trastuzumab and pertuzumab, and patients with punctate CNS haemorrhages <3 mm may be considered.

G. Prior treatment with the same class of drug unless genetic profile demonstrates a mechanism of resistance known to be potentially sensitive to trastuzumab or pertuzumab.

H. Any clinically significant concomitant disease or condition (or its treatment) that could interfere with the conduct of the trial or absorption of oral medications or that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this trial.

I. Known active infections (bacterial, fungal or viral) that would interfere with the assessment of safety or efficacy of trastuzumab and pertuzumab, including human immunodeficiency virus (HIV) positivity. Patients with history of testing positive for HIV infection are eligible provided the each of the following conditions are met:

* CD4 count ≥350/μL;
* undetectable viral load;
* receiving antiretroviral therapy (ART) that does not interact with IMP (patients should be on established ART for at least four weeks); and
* no HIV/ acquired immune deficiency syndrome (AIDS)-associated opportunistic infection in the last 12 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  An OR is defined as the confirmed occurrence of either a Complete Response (CR) or Partial Response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 criteria (or immune related [ir]-RECIST or standard imaging criteria for specific disease e.g. Response Evaluation in Neuro Oncology criteria [RANO]). In patients with leukaemia, OR will be defined as the occurrence of CR, CRi (CR incomplete neutrophil recovery) or CRp (CR with incomplete platelet recovery). The trial will report the proportion of patients with an OR and 95% credible interval.
Durable Clinical Benefit (DCB) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  DCB is defined as the absence of disease progression for at least 24 weeks from the start of trial treatment according to RECIST Version 1.1 criteria (or ir-RECIST or standard imaging criteria for specific disease e.g. RANO criteria) and, where relevant (e.g. for haematological malignancies), by standard bone marrow response assessment criteria. Alternative definitions of DCB based on different time points may be pre-specified for particular sub-cohorts if 24 weeks is not clinically relevant. The trial will report the proportion of patients with a DCB and 95% credible interval.

SECONDARY OUTCOMES:
Duration of response (DR) | Disease assessment every 2 cycles of trastuzumab and pertuzumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose for up to 2 years.
  DR is defined as the time from the date of the first confirmed CR or PR according to RECIST 1.1 or ir-RECIST or standard imaging criteria for specific disease (e.g. RANO criteria) to the date of disease progression. The trial will report the median DR and 95% credible interval.
Best percentage change in sum of target lesion / index lesion diameters (PCSD) | Disease assessment every 2 cycles of trastuzumab and pertuzumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose for up to 2 years.
  PCSD is defined as the greatest decrease or least increase in the sum of target lesion diameters (RECIST) or index lesion diameters (irRECIST) as a percentage compared to the baseline measurement. The trial will report the mean PCSD and 95% credible interval.
Time to treatment discontinuation (TTD) | From first dose of trastuzumab and pertuzumab to discontinuation of trial treatment up to 5 years.
  TTD is defined as the time from date of starting trial treatment to date of discontinuing trial treatment, in days estimated by the median of the posterior inverse gamma probability distribution. The trial will report the median TTD and 95% credible interval.
Progression-Free Survival time (PFS) | Disease assessment every 2 cycles of trastuzumab and pertuzumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose for up to 2 years.
  PFS is defined as the time from date of starting trial treatment to date of progression or date of death without a previous progression recorded estimated by the median of the posterior inverse gamma probability distribution.
Time to Progression (TTP) | Disease assessment every 2 cycles of trastuzumab and pertuzumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose for up to 2 years.
  TTP is defined as the time from date of starting trial treatment to date of progression or date of death without recorded progression censored rather than events. The trial will report the median TTP and 95% credible interval.
Growth Modulation Index (GMI) | Disease assessment every 2 cycles of trastuzumab and pertuzumab (each cycle is 21 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits are every 3 months after last dose for up to 2 years.
  GMI is defined as the ratio of TTP with the trial protocol treatment to TTP on the most recent prior line of therapy. The trial will report the mean GMI and 95% credible interval.
Overall Survival time (OS) | Time of death or up to 2 years after the EoT visit.
  OS is defined as the time from date of starting trial treatment to date of death from any cause estimated by the median of the posterior normal probability distribution.
Occurrence of at least one Suspected Unexpected Serious Adverse Reaction (SUSAR) | From the time of consent until 28 days after last dose of trastuzumab and/or pertuzumab (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  The trial will report the number of patients who experience at least one SUSAR to trastuzumab and/or pertuzumab.
Occurrence of at least one Grade 3, 4 or 5 trastuzumab and/or pertuzumab related AE | From the time of consent until 28 days after last dose of trastuzumab or pertuzumab (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  Number of patients who experience at least one trastuzumab and/or pertuzumab related Grade 3, 4 or 5 AE according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0.
EORTC-QLQ-C30 Standardised Area Under Summary Score Curve (QLQSAUC) in adult patients | QoL surveys performed prior to inclusion, every cycle (each cycle is 21 days) and at EoT visit (up to 5 years).
  For adult populations, multiple measures of Quality of Life (QoL) will be generated from patient completion of the European Organisation for Research and Treatment of Cancer QLQ-C30 (EORTC-QLQ-C30) questionnaire (15 measures). For each patient the Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean QLQSAUC and 95% credible interval.
EQ-5D Standardised Area Under Index Value Curve (EQ5DSAUC) in adult patients | QoL surveys performed prior to inclusion, every cycle (each cycle is 21 days) and at EoT visit (up to 5 years).
  For adult populations, two measures of QoL will be generated from patient completion of the EQ-5D-5L questionnaire. For each measure, scores based on responses from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean EQ5DSAUC and 95% credible interval.
Mean change from baseline in the PedsQL 4.0 Standardised Area Under total Scale Score Curve (PedsSAUC) in paediatric patients | QoL surveys performed prior to inclusion, every cycle (each cycle is 21 days) and at EoT visit (up to 5 years).
  For paediatric populations, multiple measures of QoL will be generated from patient completion of the PedsQL 4.0 (4 measures). The Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean PedsSAUC and 95% credible interval.
Mean change from baseline in the PedsQL 4.0 Standardised Area Under total Scale Score Curve (PedsSAUC) in parents of paediatric patients | QoL surveys performed prior to inclusion, every cycle (each cycle is 21 days) and at EoT visit (up to 5 years).
  For paediatric populations multiple measures of QoL will be generated from patient's parent completion of the PedsQL 4.0 (4 measures). The Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean PedsSAUC and 95% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krebs, Dr, Principal Investigator — The Christie Hospital
Locations (27):
- United Kingdom (27):
  - Belfast City Hospital, Belfast
  - University Hospital Birmingham, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Cardiff Children's Hospital, Cardiff
  - Western General Hospital, Edinburgh
  - The Beatson Hospital, Glasgow
  - Royal Hospital for Children Glasgow, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Hospital, Liverpool
  - University College London Hospital, London
  - Guy's Hospital, London
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Great North Children's Hospital, Newcastle
  - Freeman Hospital, Newcastle
  - Churchill Hospital, Oxford
  - John Radcliffe Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Sheffield's Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified patient data will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All requests for data relating to this treatment arm that are made within 5 years from last patient last visit for the trastuzumab and pertuzumab treatment arm will be considered; requests made subsequently will be considered where possible.
Access Criteria: When a request has been approved, Cancer Research UK will provide access to the de-identified individual patient-level data and appropriate supporting information. A signed Data Sharing Agreement must be in place before accessing requested information. Requests should be submitted to drugdev@cancer.org.uk.

REFERENCES:
- See also: Overview of the DETERMINE trial. — http://CRUK.org/determine
- See also: ClinicalTrials.gov record for DETERMINE Trial Master Screening Protocol (NCT05722886). — https://clinicaltrials.gov/ct2/show/NCT05722886